CLINICAL TRIAL: NCT04025827
Title: Weight Patterns in the Month After Birth: Relationship With Dietary Intake
Brief Title: Weight Patterns in the Month After Birth
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Makerere University (Other); Aga Khan University (Other); International Partnership for Human Development (Unknown); Kathmandu University School of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: A132356
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Stunting; Wasting; Undernutrition; Feeding Patterns; Feeding; Difficult, Newborn; Feeding, Breast
MeSH Terms: conditions — Growth Disorders; Cachexia; Malnutrition; Feeding Behavior; Breast Feeding | interventions — Eating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Dietary intake — We will collect detailed data on dietary intake and weight for healthy newborns in four low income countries.

SUMMARY:
This is a prospective cohort study that will be conducted in four low income countries to describe newborn weight patterns in the first month after birth and their association with clinical and demographic factors including dietary intake.

DETAILED DESCRIPTION:
Background: Worldwide, more than 50 million children under 5 are wasted (weight-for-length/height Z-score (WLZ) <-2) and over 150 million children under 5 are stunted (length/height-for-age Z-score (LAZ) <-2); such wasting and stunting often begin during infancy. Optimal early nutrition can prevent wasting and stunting. In low income countries, there is therefore a need to understand early weight patterns and how they relate to dietary intakes.

Objectives: The proposed study will assess the relationship between infant dietary intake and weight change in low income countries by characterizing neonatal weight loss/gain patterns, dietary intake, and growth.

Methodology: We will use a prospective cohort study design to describe early infant weight patterns and their relationship to dietary intake. Up to 880 newborns and their mothers will be enrolled in four countries: Guinea-Bissau, Nepal, Pakistan and Uganda (up to 220 newborns/site). Enrolled infants will be followed from birth until one month of age and will be assessed by anthropometry, dietary survey and hemoglobin measurement. Mothers will also be assessed for anthropometry and hemoglobin. Infants' fathers and next-oldest siblings will also be enrolled for anthropometry if available and willing to participate.

Descriptive statistics will be used to describe sample characteristics. We will use various regression modeling techniques to examine the links between individual, family, and community characteristics and early infant weight patterns. Logistic regression models will also be used to consider potential confounding.

Study findings will allow us to describe weight patterns in the first 30 days after birth and their relationship to the dietary intake during that time. We hypothesize that infants who lose 6% or more of their birth weight prior to beginning weight gain will have lower WAZ at 30 days of age. We also hypothesize that at 12 days of age, weight change relative to birth weight will be lower for infants born <2500g then for infants born ≥2500g.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight ≥ 2000g.
* Mother ≥18 years of age and intends to breastfeed for at least 6 months.
* Mother anticipates availability for all study visits.

Exclusion Criteria:

* Birth weight <2000g
* Respiratory distress including tachypnea, head nodding, nasal flaring, chest retractions or grunting
* Known major congenital anomalies including orofacial clefts, neural tube defects and congenital heart defects
* Contraindication to breastfeeding at each site as determined by a site's national or sub-national health authorities
* Twins and other multiples.
* Newborns whose birth weight was not obtained in the first six hours.
* Newborns whose mothers intend to move or otherwise become unavailable during the follow up period of 30 days after birth

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study will enroll singleton, healthy newborns with birth weight ≥2000 g and their mothers. Fathers and next oldest siblings also will be enrolled if available and if any indicated assent/consent is able to be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 741 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Weight for age z-score | 30 days
  Weight for age z-score
Weight change relative to birth weight | 12 days
  The difference between birth weight and current weight, expressed as a proportion of birth weight

SECONDARY OUTCOMES:
Weight equal to or exceeding birth weight | 12 days of age
  Infant weight equal to or exceeding birth weight
Weight nadir | 30 days
  Lowest weight in the first 30 days after birth, expressed as a proportion of birth weight
Age at weight nadir | 30 days
  Age in days at the time of the lowest weight in the first 30 days after birth
Weight for length z-score | 30 days
  Weight for length z-score

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flaherman, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (5):
- University of California, San Francisco, San Francisco, California, United States
- International Partnership for Human Development, Bissau, Guinea-Bissau
- Dhulikhel Hospital, Dhulikhel, Nepal
- Aga Khan University, Karachi, Pakistan
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Six months after completion of this multi-component project, unless otherwise agreed with the funder, we will make fully de-identified data from this study publicly available in a manner and under conditions agreed to by the funder, as required by the funder's Open Access Policy.
Supporting Information: Study Protocol, ICF
Time Frame: Six months after completion of the multi-component project which includes qualitative and quantitative assessment
Access Criteria: Specified by the funder's Open Access Policy

REFERENCES:
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] Aguayo VM, Menon P. Stop stunting: improving child feeding, women's nutrition and household sanitation in South Asia. Matern Child Nutr. 2016 May;12 Suppl 1(Suppl 1):3-11. doi: 10.1111/mcn.12283. PMID 27187906
- [Background] Engebretsen IM, Jackson D, Fadnes LT, Nankabirwa V, Diallo AH, Doherty T, Lombard C, Swanvelder S, Nankunda J, Ramokolo V, Sanders D, Wamani H, Meda N, Tumwine JK, Ekstrom EC, Van de Perre P, Kankasa C, Sommerfelt H, Tylleskar T; PROMISE EBF-study group. Growth effects of exclusive breastfeeding promotion by peer counsellors in sub-Saharan Africa: the cluster-randomised PROMISE EBF trial. BMC Public Health. 2014 Jun 21;14:633. doi: 10.1186/1471-2458-14-633. PMID 24950759
- [Background] Jakobsen MS, Sodemann M, Biai S, Nielsen J, Aaby P. Promotion of exclusive breastfeeding is not likely to be cost effective in West Africa. A randomized intervention study from Guinea-Bissau. Acta Paediatr. 2008 Jan;97(1):68-75. doi: 10.1111/j.1651-2227.2007.00532.x. Epub 2007 Dec 3. PMID 18053000
- [Background] Paul IM, Schaefer EW, Miller JR, Kuzniewicz MW, Li SX, Walsh EM, Flaherman VJ. Weight Change Nomograms for the First Month After Birth. Pediatrics. 2016 Dec;138(6):e20162625. doi: 10.1542/peds.2016-2625. Epub 2016 Nov 9. PMID 27940721
- [Background] Flaherman VJ, Schaefer EW, Kuzniewicz MW, Li SX, Walsh EM, Paul IM. Early weight loss nomograms for exclusively breastfed newborns. Pediatrics. 2015 Jan;135(1):e16-23. doi: 10.1542/peds.2014-1532. Epub 2014 Dec 1. PMID 25554815
- [Background] Flaherman VJ, Schaefer EW, Kuzniewicz MK, Li S, Walsh E, Paul IM. Newborn Weight Loss During Birth Hospitalization and Breastfeeding Outcomes Through Age 1 Month. J Hum Lact. 2017 Feb;33(1):225-230. doi: 10.1177/0890334416680181. Epub 2017 Jan 20. PMID 28107100